CLINICAL TRIAL: NCT00101244
Title: A Phase I, Open-Label, Dose-Escalation Study of SB-715992 Administered Days 1-3 of a 21-Day Cycle in Patients With Solid Tumors
Brief Title: SB-715992 in Treating Patients With Metastatic or Unresectable Solid Tumors or Hodgkin's or Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively Complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03193; C-2818; U01CA062487 (NIH); CDR0000404369 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — ispinesib; CK0238273

ARMS (1):
- Treatment (ispinesib) (Experimental): Patients receive SB-715992 IV over 1 hour on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of SB-715992 until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 additional patients are treated at the MTD.
  Interventions: Drug: ispinesib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: ispinesib — Given IV
  Other Names: CK0238273; SB-715992
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of SB-715992 in treating patients with metastatic or unresectable solid tumors or Hodgkin's or non-Hodgkin's lymphoma. Drugs used in chemotherapy, such as SB-715992, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of SB-715992 administered as a 1-hr intravenous infusion on days 1-3 of a 21-day cycle in patients with solid tumors.

II. To determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of SB-715992 for this administration schedule.

SECONDARY OBJECTIVES:

I. To observe clinical response of SB-715992 given days 1-3, every 21-days. II. To characterize the pharmacokinetics (PK) of SB-715992 for this administration schedule.

III. To explore drug metabolism, molecular and cellular predictors of efficacy (biomarkers) and toxicity and drug interaction potential.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive SB-715992 IV over 1 hour on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SB-715992 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 additional patients are treated at the MTD

Patients are followed for 4 weeks.

PROJECTED ACCRUAL: A total of 18-31 patients will be accrued for this study within 11-19 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; patients with solid hematologic malignancies (Hodgkin's and non-Hodgkin's lymphomas) may be included as long as a bone marrow has been performed within 6 weeks of enrollment
* Prior chemotherapy is allowed; patients may not have received chemotherapy for 4 weeks prior to the initiation of study treatment and must have full recovery from the acute effects of any prior chemotherapy; patients must not have had nitrosoureas or mitomycin C for 6 weeks prior to initiation of study treatment
* Prior radiation therapy is allowed; patients must have completed radiation at least 4 weeks prior to initiation of study treatment; patients who have received prior radiation to 50% or more of their total marrow volume will be excluded
* Prior treatment with EGFR inhibitors is allowed; prior experimental therapies (non FDA-approved agents) and immunotherapies are allowed; patients may not have received these therapies for 4 weeks prior to the initiation of study treatment and must have a full recovery from the acute effects of these therapies
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of > 12 weeks
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine =< 1.5 X institutional upper limit of normal OR creatinine clearance (calculated) or measured clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of SB-715992 on the developing human fetus are unknown; for this reason and because mitotic inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from acute AEs due to agents administered more than 4 weeks earlier
* Patients may not have received any other investigational agents within 28 days of study entry
* Patients may not receive any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) while on this study except for medications that are prescribed for supportive care but potentially may have anticancer effect (i.e. megestrol acetate, bisphosphonates); these medications must have been started 1 month prior to enrollment on study; in addition, men receiving treatment for prostate cancer will be maintained at castrate levels of testosterone by continuation of luteinizing- releasing hormone agonists
* Prohibited medications: SB-715992 is a moderate to significant in vitro inhibitor of CYP3A4; the following lists of medications/substances are moderate to significant inhibitors/inducers of CYP3A4 that, if administered concomitantly with SB-715992, may alter study drug exposure; the use of these medications/substances within 14 days (>= 6 months for amiodarone) prior to the administration of the first dose of SB-715992 through discontinuation from the study is prohibited;

  * Inhibitors of CYP3A4

    * Antibiotics: clarithromycin, erythromycin, troleandomycin
    * Antifungals: itraconazole, ketoconazole, fluconazole (doses > 200 mg/day), voriconazole
    * Antidepressants: nefazodone, fluovoxamine
    * Calcium channel blockers: verapamil, diltiazem
    * Bitter Orange
    * Miscellaneous: amiodarone*, grapefruit juice**; *use of amiodarone within 6 months prior to the administration of the first dose of SB-715992 is prohibited; ** use of grapefruit juice within 7 days prior to administration of the first dose of SB-715992 is prohibited
  * Inducers of CYP3A4

    * Anticonvulsants: phenytoin, carbamazepine, phenobarbital
    * Antibiotics: rifampin, rifabutin, rifapentine
    * Miscellaneous: St. John's wort, modafinil, oxcarbazepine
* Patients with known, symptomatic or untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because SB-715992 is a mitotic inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with SB-715992, breastfeeding should be discontinued if the mother is treated with SB-715992
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with SB-715992; appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Patients are ineligible for participation in the Drug Interaction study, or can be deemed to be ineligible to receive certain drug probes, if they have:

  * Sensitivity to sulfa drugs or adverse reactions to sulfonylureas
  * Concurrent antifungal medications, or within the past 4 weeks
  * Diabetes or other glucose imbalance
  * Acidosis
  * Concurrent alcohol use (based on the discretion of treating physician)
  * Concurrent phenytoin or diazepam treatment, or within the past 4 weeks
  * Previous intolerance to benzodiazepam therapies
  * A patient maybe excluded from all or a portion of the Drug Interaction study based on the medical discretion of the investigator
  * EVEN THOUGH PATIENTS MAY BE INELIGIBLE TO PARTICIPATE IN THE DRUG INTERACTION STUDY, THEY CAN STILL PARTICIPATE IN THE PHASE I CLINICAL TRIAL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-11; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD), based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0 | Up to 21 days

SECONDARY OUTCOMES:
Clinical response (complete response [CR], partial response [PR], and response duration) based on the Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 6 years
  Both point and confidence interval estimates of response rate will be calculated for all eligible patients (the intention to treat population), and for response-evaluable patients (the per-protocol population). Response duration will be calculated using the standard Kaplan-Meier estimator for a censored time-to-event endpoint.
Plasma ispinesib concentration levels | Up to day 24
  Descriptive statistics will be computed, including both point and confidence interval estimates.
Pre- and post-treatment intra-tumoral drug levels (from tumor-accessible, consenting patients only) | Up to day 3
  Descriptive statistics will be computed, including both point and confidence interval estimates.
Cluster of differentiation (CD)34+ stem cell levels | Pre-treatment
  Descriptive statistics will be computed, including both point and confidence interval estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States